CLINICAL TRIAL: NCT05740761
Title: Personalized MECP2 Gene Therapy Using CRISPR/Cas9 Technology Coupled to AAV-mediated Delivery in 3D Cell Culture and KI Mice
Brief Title: Gene Editing as a Therapeutic Approach for Rett Syndrome
Acronym: MECPer-3D
Status: Recruiting | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Ilaria Meloni, Associate professor, University of Siena
Other Study IDs: MECPer-3D
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — Gene Editing; In Vitro Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Gene editing in vitro — Testing of gene editing efficiency in vitro in human cellular models derived from patients

SUMMARY:
We designed the project to validate CRISPR/Cas9-based gene editing combined with AAV-based delivery for correction of the most common MECP2 mutations both in vitro and in vivo.

DETAILED DESCRIPTION:
The project aims to validate CRISPR/Cas9-based gene editing combined with AAV-based delivery for correction of the most common MECP2 mutations both in vitro and in vivo. The laboratory of the principal investigator is an active member of the European Reference Network for rare malformation syndromes and rare intellectual and neurodevelopmental disorders (ERN-ITHACA).

ELIGIBILITY:
Inclusion Criteria:

* Patients -exclusively female- since the pathology is linked to the X chromosome, with a clinical diagnosis of Rett syndrome confirmed at the genetic level by the identification, through NGS analysis, for one of the recurrent mutations (mutational hotspots) in the MECP2 gene object of the study:

  c. 473C>T - (p.(T158M)), c.502C>T (p(R168X)), c.763C>T (p.(R255X)), c.916C>T (p.(R306C));
* Age above 6 months;
* Availability of parents or legal guardians to provide free and informed consent to participate in the study

Exclusion Criteria:

* NGS diagnosis with the normal outcome;
* Positive NGS diagnosis for mutation in MECP2 but with the presence of a mutation different from those under study.
* Unwillingness of parents or legal guardians to provide free and informed consent to participate in the study;

Min Age: 6 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Rett Syndrome affects almost exclusively females
Study Population: Patients affected by Rett syndrome with one of the four hotspots mutations in MECP2 gene: p.T158M, p.R255X, p.R168X, p.R306C
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Editing efficiency | 3 years
  Percentage of gene editing achieved for each mutation

SECONDARY OUTCOMES:
Editing specificity | 3 years
  Evaluation of off-targets

CONTACTS AND LOCATIONS:
Locations (1):
- University of Siena, Siena, Siena, Italy

IPD SHARING:
Plan to Share IPD: No